CLINICAL TRIAL: NCT05338814
Title: Effects of Conventional Neck Exercise With and Without Scapular Corrective Exercises on Pain, Cervical Range of Motion and Disability in Patients With Forward Head Posture
Brief Title: Conventional Neck Exercise With and Without Scapular Corrective Exercises in Patients With Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0141 Rida
Record Dates: First submitted 2022-04-15; First posted 2022-04-21 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Forward Head Posture
Keywords: Forward head posture; Neck pain; conventional neck exercises; scapular corrective exercises
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional neck exercises & scapular corrective exercise (Experimental): isometric & stretching exercises of neck plus scapular corrective exercise
  Interventions: Other: scapular corrective exercises; Other: conventional neck exercises
- conventional neck exercises (Active Comparator): isometric & stretching exercises of neck
  Interventions: Other: conventional neck exercises

INTERVENTIONS:
Other: scapular corrective exercises — 40 minutes each, three times a week for six weeks
  Arms: conventional neck exercises & scapular corrective exercise
Other: conventional neck exercises — 40 minutes each, three times a week for six weeks

SUMMARY:
To determine the effects of conventional neck exercises with and without scapular corrective exercises on pain, cervical range of motion and disability in patients with forward head posture

ELIGIBILITY:
Inclusion Criteria:

* forward head posture
* complain of pain for at least 3months
* no history of any therapeutic interventions for the last 3months

Exclusion Criteria:

* history of whiplash injury
* any cervical surgery
* previous history of significant trauma
* fracture of cervical or scapula
* neurological impairments
* cervicogenic head ache

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 6 weeks
  it is a subjective measure in which individuals rate their pain on an eleven point numeric scale. It is composed of 0(no pain at all) to (worst imaginable pain)
Goniometry | 6 weeks
  A goniometer is a device that measures an angle or permits the rotation of anobject to a definite position
Neck disability index (NDI) | 6 weeks
  s a self-reported questionare with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation

CONTACTS AND LOCATIONS:
Overall Officials: hina gul, t-DPT, Principal Investigator — Riphah International University
Locations (1):
- Flah-e-Milat Hospital, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee K-S. Effect of a five-week scapular correction exercise in patients with chronic mechanical neck pain. The Journal of Korean Physical Therapy. 2020;32(2):126-31.
- [Background] Chen YH, Huang CY, Liang WA, Lin CR, Chao YH. Effects of Conscious Control of Scapular Orientation in Oral Cancer Survivors With Scapular Dyskinesis: A Randomized Controlled Trial. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211040827. doi: 10.1177/15347354211040827. PMID 34412536
- [Background] de Zoete RM, Brown L, Oliveira K, Penglaze L, Rex R, Sawtell B, et al. The effectiveness of general physical exercise for individuals with chronic neck pain: a systematic review of randomised controlled trials. European Journal of Physiotherapy. 2020;22(3):141-7.
- [Background] Ha SM, Kwon OY, Yi CH, Cynn HS, Weon JH, Kim TH. Effects of scapular upward rotation exercises on alignment of scapula and clavicle and strength of scapular upward rotators in subjects with scapular downward rotation syndrome. J Electromyogr Kinesiol. 2016 Feb;26:130-6. doi: 10.1016/j.jelekin.2015.12.007. Epub 2015 Dec 22. PMID 26763601
- [Background] Ozdemir F, Toy S, Kizilay F, Avci ZT, Altay Z, Colak C. Effects of scapular stabilization exercises in patients of chronic neck pain with scapular dyskinesis: A quasi-experimental study. Turk J Phys Med Rehabil. 2021 Mar 4;67(1):77-83. doi: 10.5606/tftrd.2021.6775. eCollection 2021 Mar. PMID 33948547
- [Background] Kim DH, Kim CJ, Son SM. Neck Pain in Adults with Forward Head Posture: Effects of Craniovertebral Angle and Cervical Range of Motion. Osong Public Health Res Perspect. 2018 Dec;9(6):309-313. doi: 10.24171/j.phrp.2018.9.6.04. PMID 30584494
- [Background] Mahmoud NF, Hassan KA, Abdelmajeed SF, Moustafa IM, Silva AG. The Relationship Between Forward Head Posture and Neck Pain: a Systematic Review and Meta-Analysis. Curr Rev Musculoskelet Med. 2019 Dec;12(4):562-577. doi: 10.1007/s12178-019-09594-y. PMID 31773477
- [Background] Talati D, Varadhrajulu G, Malwade M. The effect of forward head posture on spinal curvatures in healthy subjects. Asian Pacific Journal of Health Sciences. 2018;5(1):60-3.